CLINICAL TRIAL: NCT03040310
Title: Personalized Back Rx Exercise Program With Coaching, Social Support, and Sensor-assisted Assessments as a Treatment for Discogenic Low Back Pain: A Prospective Pilot Study
Brief Title: Personalized Back Rx Exercise Program as a Treatment for Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Cornell Tech (Other); UnitedHealth Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-020
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Back Rx program (Experimental): Study patients will use their smartphone apps to view their Back Rx program content, exercises, and videos.
  Interventions: Other: Back Rx program

INTERVENTIONS:
Other: Back Rx program — The Back Rx program can be viewed via a smartphone app.

SUMMARY:
The prevalence and disability associated with discogenic low back pain are significant, and there is a general lack of widely accepted conservative treatments for the condition. A majority of previous studies that have assessed the efficacy of self-directed exercise-based rehabilitation programs did not include comprehensive metrics to confirm whether participants actually participated in the exercises prescribed. In this pilot study, the investigators hope to determine whether proxies of compliance with a daily, self-directed rehabilitation program for discogenic low back pain are correlated with participant-reported improvements in pain and function. The feasibility of a mobile interface designed to help patients with chronic low back pain track the daily management of their conditions will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain with predominantly axial symptoms (axial pain > leg pain) that are exacerbated with sitting and alleviated with walking
* Persistence of symptoms for at least 3 months
* Lumbar intervertebral disc pathology evident on magnetic resonance imaging
* 18 to 65 years old
* Computer literate; have smartphone (iPhone 5S or up, Android 2.3 or up)
* English speaking

Exclusion Criteria:

* Concurrent pathology that may contribute to patients' axial low back symptoms (e.g., spondylolysis, spondylolisthesis, facet arthropathy)
* Severe lumbar disc degeneration prior to beginning Back Rx exercise program
* History of lumbar spine surgery or other interventions prior to beginning Back Rx exercise program
* History of trauma
* Cases involving workers' compensation or other legal claims
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | Up to 12 months post-program start
  The Oswestry Disability Index is scored on a scale of 0-100, with a higher number representing more severe disability.

SECONDARY OUTCOMES:
Compliance with app/program | Up to 12 months post-program start
  Measured via usage analytics by a composite index based on % of videos viewed and % of videos completed
Satisfaction with program | Up to 12 months post-program start
  Participants will be asked whether they would recommend the app to a friend.
Medication utilization | Up to 3 months post-program start
  Usage of medications will be documented
Pain score | Up to 12 months post-program start
  Pain will be assessed via the visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Vad VB, Madrazo-Ibarra A, Estrin D, Pollak JP, Carroll KM, Vojta D, Vad A, Trapness C. "Back Rx, a personalized mobile phone application for discogenic chronic low back pain: a prospective pilot study". BMC Musculoskelet Disord. 2022 Oct 19;23(1):923. doi: 10.1186/s12891-022-05883-9. PMID 36261825
- [Derived] Selter A, Tsangouri C, Ali SB, Freed D, Vatchinsky A, Kizer J, Sahuguet A, Vojta D, Vad V, Pollak JP, Estrin D. An mHealth App for Self-Management of Chronic Lower Back Pain (Limbr): Pilot Study. JMIR Mhealth Uhealth. 2018 Sep 17;6(9):e179. doi: 10.2196/mhealth.8256. PMID 30224333